CLINICAL TRIAL: NCT02901808
Title: Interdisciplinary Retrospective Registeranalysis for the Examination of Non-occlusive Mesenteric Ischemia (NOMI)
Brief Title: Registeranalysis for the Examination of NOMI
Acronym: IRRE NOMI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Peter Minko, Assistant Medical Director, Universität des Saarlandes
Other Study IDs: 209/15
Record Dates: First submitted 2016-08-18; First posted 2016-09-15 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Mesenteric Ischemia
Keywords: NOMI; Angiography; Digital Subtraction Angiography (DSA)
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NOMI: Patients suffering from NOMI
- No-NOMI: Patients not suffering from NOMI

SUMMARY:
The registry includes patients undergoing cardiovascular and thoracic surgery at the Saarland University Medical Center, Homburg/Saar, Germany. This study is a monocentric, retrospective study investigating the development of NOMI and outcome of patients.

DETAILED DESCRIPTION:
All data were acquired from the hospital electronic health record and the picture archiving computer system (PACS).

NOMI was suspected if the following clinical signs occured:

new onset of oliguria (urine output <0.5 mL/kg/hour for at least 6 hours) or anuria, abdominal distention with decreased or absent bowel sounds, elevated serum lactate levels >5.0mmol/L or metabolic acidosis (base excess <-5mmol/L).

In accordance to the definition of cardiogenic shock angiography was performed in patients with a systolic blood pressure >90 mmHg and a cardiac index >1.8 L/minute/m².

ELIGIBILITY:
Inclusion Criteria:

* The investigators include anonymous data from patients with cardio-thoracic surgery

Exclusion Criteria:

* None

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardio-thoracic surgical patients
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2008-01; Primary Completion 2014-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Development of NOMI | at the day of surgery, day zero
  Clinical signs of NOMI

SECONDARY OUTCOMES:
Length of stay | at the day of surgery, day zero up to 365 days
  Length of stay will be measured upon the time spent on intensive care unit and in the hospital
Mechanical ventilation | at the day of surgery, day zero up to 365 days
  Length of mechanical ventilation will be measured upon the time spent on intensive care unit
Mortality | at the day of surgery, day zero up to 365 days
  Mortality will be measured upon patients leaving the hospital dead or alive.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Buecker, MD, Study Director — Department of Diagnostic and Interventional Radiology; Hans-Joachim Schäfers, MD, Study Director — Department of Thoracic and Cardiovascular Surgery
Locations (1):
- Saarland University Medical Center, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No